CLINICAL TRIAL: NCT00003602
Title: A Randomised Study Comparing an Oral Regimen (Idarubicin and Etoposide) With an Intravenous Regimen (MAE) for Consolidation in Patients Over 55 Years With Acute Myeloid Leukaemia in First Complete Remission
Brief Title: Combination Chemotherapy in Treating Older Patients With Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Riverside Haematology Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066675; RHG-AML97; EU-98031
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-01

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: untreated adult acute myeloid leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts | interventions — Cytarabine; Etoposide; Idarubicin; Mitoxantrone

INTERVENTIONS:
Drug: cytarabine
Drug: etoposide
Drug: idarubicin
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating older patients with acute myeloid leukemia.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different combination chemotherapy regimens in treating older patients with acute myeloid leukemia in first remission.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of oral idarubicin and etoposide vs intravenous mitoxantrone, etoposide, and cytarabine as consolidation therapy in patients over 55 years old with acute myeloid leukemia in first complete remission.
* Compare the toxicity of these 2 regimens in these patients.
* Assess the quality of life of these patients.

OUTLINE: This is a randomized study. Patients are stratified according to number of courses of induction therapy required to achieve complete remission.

All patients receive induction chemotherapy consisting of idarubicin IV on days 1-3 and cytarabine IV over 12 hours on days 1-7. Patients receive 1-2 courses of induction chemotherapy to achieve complete remission.

Patients are randomized to one of two treatment arms for consolidation therapy after achieving complete remission.

* Arm I: Patients receive 2 courses of mitoxantrone IV on days 1 and 2, etoposide IV over 1 hour on days 1-5, and cytarabine IV over 12 hours on days 1-5.
* Arm II: Patients receive 2 courses of oral idarubicin and etoposide on days 1-3.

Quality of life is assessed before each course of consolidation chemotherapy and 6-8 weeks after completion of therapy.

Patients are followed until death.

PROJECTED ACCRUAL: Approximately 400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed de novo or secondary acute myeloid leukemia (AML)

  * Prior myelodysplasia allowed
  * Refractory anemia with excess blasts (RAEB) OR
  * RAEB in transformation
* No relapsed AML
* No chronic granulocytic leukemia in transformation
* No CNS disease

PATIENT CHARACTERISTICS:

Age:

* Over 55

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Transaminases no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 2.5 times ULN

Cardiovascular:

* No severe or uncontrolled cardiac failure

Other:

* No serious medical, social, or psychological condition
* Not HIV 1 or 2 seropositive

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No plan for future autograft

Chemotherapy:

* No prior chemotherapy for myelodysplastic syndrome or AML

Endocrine therapy:

* Not specifed

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent aluminum or magnesium-based antacids

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 1998-03

CONTACTS AND LOCATIONS:
Overall Officials: Graham Jackson, MD, Study Chair — Newcastle-upon-Tyne Hospitals NHS Trust
Locations (1):
- Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England, United Kingdom